CLINICAL TRIAL: NCT03896191
Title: The Association of Gait Kinematics, Instability and Patient Reported Outcomes in Patients With Total Knee Replacement
Status: Completed | Type: Observational
Sponsor: University of Bath (Other)
Collaborators: North Bristol NHS Trust (Other)
Responsible Party: Principal Investigator, David Bruce, Principal Investigator, University of Bath
Other Study IDs: 19-03607
Record Dates: First submitted 2019-03-26; First posted 2019-03-29 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Total knee replacement; Revision knee surgery; Knee instability; Gait analysis; Patient reported outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stable, satisfied primary TKR: Participants who have a stable TKR (as assessed by the surgical team) and are satisfied with their knee replacement (as assessed by a questionnaire).
  Interventions: Other: No intervention.
- Unstable, dissatisfied primary TKR: Participants who are dissatisfied with their TKR, with instability (including instability due to aseptic loosening) and consequently awaiting revision TKR.
  Interventions: Procedure: Revision TKR surgery

INTERVENTIONS:
Procedure: Revision TKR surgery — This study will follow the cohort of patients who have an unstable primary TKR with which they are dissatisfied. They will be assessed before and after their revision TKR surgery.
  Groups: Unstable, dissatisfied primary TKR
Other: No intervention. — This study will also make a case-control comparison between patients with a stable primary TKR and an unstable primary TKR.
  Groups: Stable, satisfied primary TKR

SUMMARY:
It is unclear why 20% of patients with total knee replacements (TKR) are dissatisfied. Few studies have specifically assessed the way people walk ('gait') with an 'unhappy' or unstable knee or following re-do ('revision') TKR surgery.

The investigators conjecture that people having re-do TKR surgery because their knee is unstable will have altered walking patterns (for example, less bending of the knee) before and after surgery, and that these changes are related to how satisfied the patient is with their knee. The investigators will also examine whether there are differences in the way people walk with an unstable knee replacement or with a stable knee replacement, in comparison to people who do not have a knee replacement.

This exploratory project will use 3D infrared cameras to analyse differences in walking patterns and whether there is associated change in patient satisfaction. If an association exists, the data from this study may help to develop alternative measures of outcomes, in order to guide treatment decisions.

DETAILED DESCRIPTION:
The effect of TKR instability on gait is poorly understood. How does revision TKR surgery for instability alter gait and is there an associated change in patient satisfaction? Are there differences in gait between patients with an unstable TKR and a stable TKR? The objectives of this study are:

1. To investigate the effect of a revision TKR operation on gait kinematics, in patients who have a primary TKR and instability.
2. To investigate the association between changes in gait kinematics and patient satisfaction, before and after revision TKR surgery for patients with instability.
3. To investigate differences in gait kinematics between dissatisfied patients with an unstable primary TKR, satisfied patients with a stable primary TKR and people who do not have a knee replacement.

The first part of the investigation will tackle the first two objectives and follow patients who are having a revision TKR due to an unstable knee before and after their operation. The second part will then compare these patients to those with a primary TKR and no instability and to a control group of participants who do not have knee replacements ('native knees') and do not have difficulty walking. This will determine the difference in kinematics between a native knee and a TKR with and without instability.

Age, height, weight, leg lengths, measurements of the TKR position on imaging (taken as part of routine clinical practice) and patient reported outcome scores will be documented.

The gait assessments will be carried out in the outpatient clinic or physiotherapy department. These patients will have their walking gait assessed using a treadmill-based portable 3D infrared camera system (Vicon Ltd, Oxford, UK). The raw data will be processed by Run3D (Run3D Ltd, Oxford, UK) and Visual3D (C-motion Inc, MD, USA) to calculate knee joint angles.

Analysis will focus on within subject (part 1) and between subject differences (part 2). The questions are novel and data will be largely exploratory. Measures, differences and correlations will be presented using descriptive statistics and, where appropriate, correlation and regression coefficients. Where possible, inferential statistics (such as t-tests) will formally test differences in knee kinematic measures and associations with PROMS. Statistical parametric mapping will be applied to analyse continuous quantities over the gait cycle. Published research indicates an effect size of 1.0 may be expected. This suggests sample sizes between 11 and 42 should be sufficient to determine statistically significant two-tailed differences (alpha=0.05, beta=0.2) within subjects or between groups, according to the comparison being assessed. A sample of 42 patients is targeted.

In the longer term, this study will enable a better understanding of the functional biomechanics of TKR instability and potentially develop an alternative quantitative measurement of outcome and instability.

ELIGIBILITY:
Inclusion Criteria:

Patients awaiting revision TKR due to instability:

* Patients who have a primary total knee replacement.
* Patients who have an unstable knee replacement, as determined by the surgical team.
* Patients who are being listed for a revision total knee replacement.

Primary TKR without instability:

* Patients with a primary total knee replacement.
* Patients at least one year after their primary total knee replacement operation.

Exclusion Criteria:

Patients awaiting revision TKR due to instability:

* Patients who have suspected infection of the TKR.
* Patients who are awaiting a two-stage revision procedure.
* Patients who can walk less than one minute at a time.
* Patients who can walk for less than five minutes with rests.
* Patient who are not able to give informed consent.

Primary TKR without instability:

* Patients who have had a previous revision of the total knee replacement.
* Patients who have an unstable knee replacement, as determined by the surgical team.
* Patients who have aseptic loosening or wear, as determined by the surgical team.
* Patients who are not satisfied with their TKR (as determined by the study specific questionnaire).
* Patients who can walk for less than one minute at a time.
* Patients who can walk for less than five minutes with rests.
* Patient who are not able to give informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending orthopaedic knee clincs at a tertiary referral hospital.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Change from preoperative maximum knee flexion during swing. | 8-12 weeks after surgery.
  Maximum knee flexion angle during the swing phase of gait.
Change from preoperative maximum knee flexion during swing. | 1 year after surgery.
  Maximum knee flexion angle during the swing phase of gait.

SECONDARY OUTCOMES:
Change from preoperative maximum knee flexion during stance. | 8-12 weeks after surgery.
  Maximum knee flexion angle during the stance phase of gait.
Change from preoperative maximum knee flexion during stance. | 1 year after surgery.
  Maximum knee flexion angle during the stance phase of gait.
Change from preoperative knee sagittal plane range of movement. | 8-12 weeks after surgery.
  Knee sagittal plane range of movement during stance and swing phases of gait.
Change from preoperative knee sagittal plane range of movement. | 1 year after surgery.
  Knee sagittal plane range of movement during stance and swing phases of gait.
Change from preoperative knee coronal plane range of movement. | 8-12 weeks after surgery.
  Knee coronal plane range of movement during stance and swing phases of gait.
Change from preoperative knee coronal plane range of movement. | 1 year after surgery.
  Knee coronal plane range of movement during stance and swing phases of gait.
Change from preoperative knee axial plane range of movement. | 8-12 weeks after surgery.
  Knee axial plane range of movement during stance and swing phases of gait.
Change from preoperative knee axial plane range of movement. | 1 year after surgery.
  Knee axial plane range of movement during stance and swing phases of gait.
Change from preoperative baseline in Oxford Knee Score. | 8-12 weeks after surgery.
  Patient reported outcome measure. Minimum 0, Maximum 48 (48 being best).
Change from preoperative baseline in Oxford Knee Score. | 1 year after surgery.
  Patient reported outcome measure. Minimum 0, Maximum 48 (48 being best).
Change from preoperative baseline in Knee injury and Osteoarthritis Outcome Score. | 8-12 weeks after surgery.
  Patient reported outcome measure. Minimum 0, Maximum 100 (100 being best). Subscales (pain, symptoms, function, sports and recreation, quality of life) are transformed to the 0-100 overall scale.
Change from preoperative baseline in Knee injury and Osteoarthritis Outcome Score. | 1 year after surgery.
  Patient reported outcome measure. Minimum 0, Maximum 100 (100 being best). Subscales (pain, symptoms, function, sports and recreation, quality of life) are transformed to the 0-100 overall scale.
Change from preoperative baseline in American Knee Society Score. | 8-12 weeks after surgery.
  Patient reported outcome measure with two subscales. Subscales are the Knee Society Score, Minimum 0, Maximum 100 (100 being best); and Knee Society Function Score Minimum 0, Maximum 100 (100 being best).
Change from preoperative baseline in American Knee Society Score. | 1 year after surgery.
  Patient reported outcome measure with two subscales. Subscales are the Knee Society Score, Minimum 0, Maximum 100 (100 being best); and Knee Society Function Score Minimum 0, Maximum 100 (100 being best).
Change from preoperative baseline in EQ-5D-5L questionnaire. | 8-12 weeks after surgery.
  Patient reported outcome measure. Subcategories (mobility, self-care, activity, pain, anxiety) scored between 1 and 5 (1 being best) and a visual analog score between 0 and 100 (100 being best).
Change from preoperative baseline in EQ-5D-5L questionnaire. | 1 year after surgery.
  Patient reported outcome measure. Subcategories (mobility, self-care, activity, pain, anxiety) scored between 1 and 5 (1 being best) and a visual analog score between 0 and 100 (100 being best).

OTHER OUTCOMES:
Statistical parametric mapping of sagittal plane knee kinematics. | 8-12 weeks after surgery.
  Analysis of the whole gait cycle compared to preoperative kinematics.
Statistical parametric mapping of sagittal plane knee kinematics. | 1 year after surgery.
  Analysis of the whole gait cycle compared to preoperative kinematics.
Statistical parametric mapping of coronal plane knee kinematics. | 8-12 weeks after surgery.
  Analysis of the whole gait cycle compared to preoperative kinematics.
Statistical parametric mapping of coronal plane knee kinematics. | 1 year after surgery.
  Analysis of the whole gait cycle compared to preoperative kinematics.
Statistical parametric mapping of axial plane knee kinematics. | 8-12 weeks after surgery.
  Analysis of the whole gait cycle compared to preoperative kinematics.
Statistical parametric mapping of axial plane knee kinematics. | 1 year after surgery.
  Analysis of the whole gait cycle compared to preoperative kinematics.
Variability of the primary and secondary outcome measures outlined above. | 8-12 weeks after surgery.
  Variability compared to preoperative kinematics.
Variability of the primary and secondary outcome measures outlined above. | 1 year after surgery.
  Variability compared to preoperative kinematics.
The above outcomes will also be applied to the hip and ankle joints. | 8-12 weeks after surgery.
  These comparisons will assess change compared to preoperative kinematics.
The above outcomes will also be applied to the hip and ankle joints. | 1 year after surgery.
  These comparisons will assess change compared to preoperative kinematics.

CONTACTS AND LOCATIONS:
Overall Officials: David J Bruce, BA, BMBCh, Principal Investigator — University of Bath
Locations (1):
- Southmead Hospital, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The final anonymised raw and processed datasets will be made available for future research, as specified in the University of Bath's data management guidelines.
Supporting Information: Study Protocol, CSR
Time Frame: Anonymised data will be made openly available to other researchers one year after completion of the study, or from the first publication using data from the study. The data will be stored on the Bath research archive for a period of at least 10 years.
Access Criteria: Anonymised data will be made available to bona fide researchers who will need to request access via the University of Bath research archive (https://researchdata.bath.ac.uk/).